CLINICAL TRIAL: NCT01634074
Title: A Multicenter, Prospective, Variable Duration, Reiterative Development and Evaluation Study of ApniCure's Therapy System(s) for the Treatment of Obstructive Sleep Apnea (OSA)
Brief Title: Reiterative Development and Evaluation Study of OSA Therapy System
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: ApniCure, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: 11847
Record Dates: First submitted 2012-07-03; First posted 2012-07-06 (Estimated); Last update posted 2013-11-25 (Estimated); Status verified 2013-11

CONDITIONS: Obstructive Sleep Apnea
MeSH Terms: conditions — Sleep Apnea, Obstructive

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- OSA patients: Patients with Obstructive Sleep Apnea (OSA), or suspected OSA

SUMMARY:
The purpose of this study is to evaluate new iterations/generations of the ApniCure sleep therapy device.

ELIGIBILITY:
Inclusion Criteria:

1. Subject is between the ages of 18 and 80.
2. Subject is fluent in English and understands the Study protocol and is willing and able to comply with Study requirements and sign the informed consent form.
3. Subject has a least one molar in each of the four quadrants of the mouth (right upper, right lower, left upper, and left lower).

Exclusion Criteria:

1. Poor nasal patency as evidenced by the inability to breathe through the nose with the mouth closed.
2. Oral cavity infection or any other oral or dental condition or problem that would limit subject use of the ApniCure System (e.g. dentures, loose tooth/teeth, temporomandibular joint (TMJ) conditions, or any oral or dental condition that the Investigator believes could be exacerbated by the Attune Sleep Apnea System.
3. History of any OSA surgical treatment including uvulopalatopharyngoplasty surgery (UPPP), maxillomandibular advancement surgery (MMA), radio frequency (RF) ablation treatment, palatal stent devices, etc.
4. Any concomitant diagnosed or suspected sleep or chronic neurological disorders, other than OSA, including insomnia, and central sleep apnea.
5. Currently working nights, or rotating night shifts.
6. Current disease state, use of medication or other treatment which, in the investigator's opinion, may pose additional risk to the subject or confound the results of the study.
7. Female subjects of child bearing age who are pregnant or intend to become pregnant during the study period.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with known or suspected OSA
Sampling Method: Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2012-07; Primary Completion 2014-07 (Estimated); Study Completion 2014-07 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Mehran Farid-Moayer, MD, Principal Investigator — Peninsula Sleep lab
Locations (7):
- United States (7):
  - Penninsula Sleep Center (PSC), Burlingame, California
  - ApniCure, Inc., Redwood City, California
  - Sleep Disorders Center of Georgia (SDCG), Atlanta, Georgia
  - Kentucky Research Group, Louisville, Kentucky
  - The Center for Sleep & Wake Disorders, Chevy Chase, Maryland
  - SleepMed, Columbia, South Carolina
  - Sleep Medicine Associates of Texas (SMAT), Dallas, Texas